CLINICAL TRIAL: NCT03190993
Title: The Diet Composition and Energy Balance Pilot Study
Brief Title: The DEB Pilot Study
Acronym: DEB Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual); Owen T. Carmichael (Unknown)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6218
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Nutritional Physiological Phenomena; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A randomized parallel arm design trial examining solid sugar vs. SSB treatments will be performed.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar Sweetened Solid Treatment (Active Comparator): A solidified food that is made with the SSB syrup concentrate and gelatin. It is equivalent to one 20 oz. soft drink.
  Interventions: Other: Sugar Sweetened Solid Treatment
- Sugar Sweetened Beverage Treatment (Active Comparator): 20 oz. carbonated sugar sweetened beverage. Added ingredients include: ~2.1g whey protein powder.
  Interventions: Other: Sugar Sweetened Beverage Treatment

INTERVENTIONS:
Other: Sugar Sweetened Solid Treatment — Consume Sugar Sweetened Solid Treatment (product) daily.
  Arms: Sugar Sweetened Solid Treatment
Other: Sugar Sweetened Beverage Treatment — Consume Sugar Sweetened Beverage Treatment (product) daily.
  Other Names: SSB Treatment
  Arms: Sugar Sweetened Beverage Treatment

SUMMARY:
The purpose of the current study is to test if weight change is differentially affected by consumption of foods that are identical in carbohydrate (i.e. sugar) but vary in food form over 1 month.

DETAILED DESCRIPTION:
Dose: Participants are to consume 1 unit per day of the study product.

Diet: Participants will receive no instructions for other dietary modifications; i.e., they will not be told to modify what or how much other food they consume.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20 - 40

Exclusion Criteria:

* Diabetes (Type 1 or 2)
* Prediabetes
* Active cancer
* Serious digestive disorders
* Other conditions that affect metabolism or body weight
* Uncontrolled Thyroid disorder (controlled = 6 months of medication)
* Unable to consume study foods
* Non- weight stable (more than 10 lbs weight gain or loss in last 6 months)
* Pregnancy
* Intentions of becoming pregnant in the next 2 months
* Women who have undergone partial hysterectomy with intact ovary function
* Current or past alcohol or drug abuse problem
* Allergy or intolerance to study product ingredients.
* Any other medical, psychiatric or behavioral factors that in the judgment of the Principle Investigator that may interfere with study participation or the ability to follow the protocol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Sweetened Solid Treatment | Sugar Sweetened Beverage Treatment
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Sweetened Solid Treatment | Sugar Sweetened Beverage Treatment | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 36 [21 to 50] | 39 [25 to 56] | 37 [21 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight at 1 month
Time Frame: 1 month
Measure: Mean (Standard Error); unit: kg
Arm/Group | Sugar Sweetened Solid Treatment | Sugar Sweetened Beverage Treatment
Number analyzed (Participants) | 10 | 10
kg | -0.325 (0.307) | 0.230 (0.307)
Statistical Analysis 1: Comparison: Sugar Sweetened Solid Treatment vs Sugar Sweetened Beverage Treatment; Test type: Other — Linear mixed effect models were used to test if changes (Day 28 - Baseline) were equal between treatment groups (primary outcome); p = 0.22, Regression, Linear; Mean Difference (Net) = 0.56, Standard Error of Mean 0.43

ADVERSE EVENTS:
Time Frame: 4 weeks.
Arm/Group | Sugar Sweetened Solid Treatment | Sugar Sweetened Beverage Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT03190993/ICF_000.pdf
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT03190993/Prot_001.pdf